CLINICAL TRIAL: NCT02467075
Title: Phase IV Randomized Double-Blinded Placebo-Controlled Noninferiority Study of the Effect of Intravenous Low-Osmolality Iodinated Contrast Material On Renal Function in Postoperative Adults With Stage IIIb or Stage IV Chronic Kidney Disease
Brief Title: Double-Blind Placebo-Controlled CIN Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient number of subjects could be enrolled.
Sponsor: University of Michigan (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Matthew Davenport, MD, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HUM 00097944
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Acute Kidney Injury
Keywords: CT, iodinated contrast, contrast-induced AKI, kidney injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Contrast Media; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Iopamidol 300 (Contrast) (Active Comparator): Subjects scheduled for a clinical CT will be randomized to receive weight-based low-osmolality iodinated contrast with the CT. All subjects will receive a minimum of 1 mL/kg/hr of isotonic volume expansion for at least three hours before and three hours after the CT.
  Interventions: Drug: Iopamidol 300 (Contrast)
- Placebo (Normal Saline) (Placebo Comparator): Subjects scheduled for a standard of care CT will be randomized to receive weight-based normal saline instead of contrast material with the CT. All subjects will receive a minimum of 1 mL/kg/hr of isotonic volume expansion for at least three hours before and three hours after the CT.
  Interventions: Drug: Placebo (Normal Saline)

INTERVENTIONS:
Drug: Iopamidol 300 (Contrast) — Patients will be randomized to receive IV iopamidol 300 (1.25 mL/kg, max 125 mL) with their CT scan
  Arms: Iopamidol 300 (Contrast)
Drug: Placebo (Normal Saline) — Patients will be randomized to receive IV normal saline (1.25 mL/kg, max 125 mL) with their CT scan
  Other Names: Normal saline
  Arms: Placebo (Normal Saline)

SUMMARY:
This double-blinded placebo-controlled study will examine the incidence and significance of contrast-induced acute kidney injury following IV iodine-based contrast material administration in subjects with stage IIIB or stage IV chronic kidney disease.

Subjects will be scheduled for clinically indicated CT of the abdomen and/or pelvis to evaluate for suspected intra-abdominal infection. Subjects will be randomized to receive either weight-based low-osmolality iodinated contrast material or saline. The primary outcome measure will be the incidence of stage II AKI by AKIN (Acute Kidney Injury Network) criteria.

DETAILED DESCRIPTION:
This double-blinded placebo-controlled non-inferiority study will examine the incidence and significance of contrast-induced acute kidney injury following intravenous iodine-based contrast material administration in subjects with stage IIIB or stage IV chronic kidney disease.

Subjects will be scheduled for clinically indicated CT of the abdomen and/or pelvis to evaluate for suspected intra-abdominal infection. Subjects will be randomized to receive either weight-based low-osmolality iodinated contrast material or saline. The primary outcome measure will be the incidence of stage II AKI by AKIN criteria.

Secondary outcome measures will include AKI by other definitions (stage I AKI, traditional CI-AKI definition), hospital length of stay, 30-day readmission rate, number of additional percutaneous interventions within 30 days, number of additional CT examinations within 30 days, and 30-day mortality rate. All subjects will receive a minimum of 1 mL/kg/hr (max: 125 mL/hr) of volume expansion for at least three hours before and after the CT..

ELIGIBILITY:
Inclusion Criteria:

* Inpatients scheduled for CT scan of abdomen and/or pelvis
* Had surgery in the last 4 weeks
* Stable renal function (based on serum creatinine-last two lab values +/- 0.3 of each other, with most recent within 5 days of CT)
* Suspected infection or fluid collection in abdomen and/or pelvis

Exclusion Criteria:

* Pregnant
* Severe Allergy (anaphylaxis) to contrast
* Dialysis in last 7 days
* Received intravascular iodinated contrast in last 48 hours
* CT of abdomen and pelvis in last 7 days shows no fluid collection
* Prisoners
* CT ordered for an indication that requires (eg, CT angiogram) or contraindicates (eg, renal stone CT) the administration of intravascular contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davenport, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital Department of Radiology, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from inpatients at a tertiary medical center who were scheduled to have a clinical CT for a suspected infection. Subjects had to have a previous diagnosis of Chronic Kidney Disease (CKD) Stage II or IIB and stable creatinine levels. Their physician had to agree to their participation in the study.
Pre-assignment Details: Patients had to be scheduled for a CT that did not have a) requirement for the CT scan to be performed with contrast agent or b) a contraindication against having the CT scan with contrast agent
Groups:
- Iopamidol 300 (Contrast): Subjects scheduled for a clinical CT will be randomized to receive weight-based low-osmolality iodinated contrast with the CT. All subjects will receive a minimum of 1 mL/kg/hr of isotonic volume expansion for at least 3 hours before and 3 hours after the CT. The function of the fluids is to minimize the effect of the contrast on their creatinine level.
  Iopamidol 300 (Contrast): Patients will be randomized to receive IV iopamidol 300 (1.25 mL/kg, up to a max volume of 125 mL) with their CT scan
- Placebo (Normal Saline): Subjects scheduled for a clinical CT will be randomized to receive normal saline instead of contrast material with the CT. All subjects will receive a minimum of 1 mL/kg/hr of isotonic volume expansion for at least 3 hours before and 3 hours after the CT. The fluids are given to placebo patients in order to minimize any differences in treatment between the treatment and placebo groups.
  Placebo (Normal Saline): Patients will be randomized to receive IV normal saline (1.25 mL/kg, up to a max volume of 125 mL) with their CT scan
Period: Initial CT Scan
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0
Period: 48 Hour Follow-up
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0
Period: 72 Hour Follow-up
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0
Period: 30 Day Follow-up
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] |  | 84 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants With Stage II AKI (Acute Kidney Injury)
Description: Participants who had Stage II AKI. This is measured by comparing an initial blood creatinine level with the level at 48 hours. Creatine is a chemical waste product that passes through the kidneys. Creatinine levels reflect how well the kidneys are working.
Time Frame: 48 hours
Population: Participants with State II AKI (Acute Kidney Injury)
Measure: Count of Participants; unit: Participants
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Number analyzed (Participants) | 0 | 1
Participants | 0 | 0

2. Secondary Outcome: Subjects With AKI (Acute Kidney Injury), Stage 1 or Other Definition
Description: Stage I AKI, traditional CIN definitions or other definitions of AKI (acute kidney injury) at lower levels of severity
Time Frame: 48-72 hours
Measure: Count of Participants; unit: Participants
Groups:
- Iopamidol 300 (Contrast): Subjects scheduled for a clinical CT were randomized to receive weight-based low-osmolality iodinated contrast with the CT.
  All subjects will receive a minimum of 1 mL/kg/hr of isotonic volume expansion for at least 3 hours before and 3 hours after the CT.
  Iopamidol 300 (Contrast): Patients will be randomized to receive IV iopamidol 300 (1.25 mL/kg, up to a max volume of 125 mL) with their CT scan
- Placebo (Normal Saline): Subjects scheduled for a clinical CT were randomized to receive weight-based normal saline instead of contrast material with the CT.
  All subjects will receive a minimum of 1 mL/kg/hr of isotonic volume expansion for at least 3 hours before and 3 hours after the CT.
  Placebo (Normal Saline): Patients will be randomized to receive IV normal saline (1.25 mL/kg, up to a max volume of 125 mL) with their CT scan
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Number analyzed (Participants) | 0 | 1
Participants | 0 | 0

3. Secondary Outcome: Subjects Requiring Renal Replacement Therapy (Kidney Transplant or Dialysis)
Description: Number of subjects that require renal (kidney) replacement therapy, such as a kidney transplant or dialysis within 30 days of study participation.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Number analyzed (Participants) | 0 | 1
Participants | 0 | 0

4. Secondary Outcome: Hospital Length of Stay
Description: Subject's hospital length of stay in days
Time Frame: Duration of hospital stay (assessed from date of randomization up to 30 days)
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: days
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Number analyzed (Participants) | 0 | 1
Number analyzed (days) | 0 | 1
days |  | 30 (0)

5. Secondary Outcome: 30-day Readmission
Description: Number of times a subject is readmitted within 30 days of study recruitment
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Number of admissions
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Number analyzed (Participants) | 0 | 1
Number of admissions |  | 0 (0)

6. Secondary Outcome: Mortality Rate - 30 Day
Description: Number of subjects who died within 30 days of entry into the study.
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
Number analyzed (Participants) | 0 | 1
participants |  | 0

ADVERSE EVENTS:
Time Frame: Subjects were followed for 30 days
Description: The same definitions of adverse events and serious adverse events has been used.
Arm/Group | Iopamidol 300 (Contrast) | Placebo (Normal Saline)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
The decision to terminate the study due to low accrual potential was made in February 2016, but last data collection from the 1 subject was in September 2015.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No